CLINICAL TRIAL: NCT01552239
Title: Phase II Study of Preoperative Radiotherapy for Sarcomas of the Extremities With Intensity-Modulation, Image-Guidance, Small Safety-margins and Brachytherapy Conditioned by Resection Margin
Brief Title: Preoperative Radiotherapy for Sarcomas of the Extremities With Intensity-Modulation, Image-Guidance and Small Safety-margins
Acronym: PREMISS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRE-1205-ROE-0050-I; No. 2009.906.1 (Other Grant/Funding Number: Wilhelm-Sander-Stiftung)
Record Dates: First submitted 2011-07-26; First posted 2012-03-13 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Soft Tissue Sarcoma of the Limb; AJCC Stage II and III
Keywords: Soft tissue sarcoma; Intensity-Modulated Radiation Therapy (IMRT); Tomotherapy; Safety Margins; Image-guided Radiation Therapy; Brachytherapy; interstitial
MeSH Terms: conditions — Sarcoma | interventions — Brachytherapy

ARMS (1):
- 1 Arm (Experimental): Stratum A:
  R0, primary wound closure
  Stratum B:
  R0, secondary wound closure
  Stratum C:
  R1, tertiary wound closure
  Interventions: Radiation: IMRT/IGRT, Tumor resection, Brachytherapy

INTERVENTIONS:
Radiation: IMRT/IGRT, Tumor resection, Brachytherapy — All:
  Preoperative IMRT with small safety margins (GTV according to MRT plus 1.5cm laterally / 3cm proximodistally) to 50Gy total dose, 2 Gy single dose, 5 fractions per week, daily IGRT with in-room CT (Tomotherapy)
  Tumor resection after 4-6 weeks
  Stratum C: Interstitial Brachytherapy to tumor bed with 15 Gy total dose, 3 Gy single dose b.i.d. in second week after tumor resection

SUMMARY:
RATIONALE: Modern radiotherapy techniques in a neoadjuvant setting have the potential to minimize morbidity and maximize efficacy. An additional boost dose can be provided locally by HDR-brachytherapy in patients with positive margins after tumor resection.

PURPOSE: This phase II trial is studying the safety and efficacy of a combination of modern radiotherapy elements applied to the tumor and small volumes of surrounding normal tissue (IMRT, IGRT; brachytherapy in case of positive resection margin) and see how well it works in treating patients with High-Risk Soft Tissue Sarcoma of the Extremities.

ELIGIBILITY:
Inclusion Criteria:

Histologic and radiographic proof of localized high-risk soft tissue sarcoma meeting the following criteria:

* Lesion originates in extremity

  * upper extremity lesions may occur from the medial border of the scapula to tumors as far distal as the finger tips
  * lower extremity regions include hip girdle tumors commencing at the iliac crest, excluding lesions arising from within the pelvis, and extends to include lesions as far distal as the toes
* AJCC Stage II or III disease (except T1a-tumors or N1)
* Primary presentation or local recurrence
* after biopsy or inadequate surgery resulting in residual tumor in cross-sectional imaging
* Tumors must be considered resectable according to cross sectional imaging, or potentially resectable after preoperative radiotherapy
* ECOG Performance Status 0-2
* Informed Consent

Exclusion Criteria:

* Diagnosis of the following:

  * Primitive neuroectodermal tumor
  * Soft tissue Ewing's sarcoma
  * Extraskeletal osteo- or chondrosarcoma
  * Aggressive fibromatosis (desmoid tumors)
  * Dermatofibrosarcoma protuberans
* Regional nodal disease or unequivocal distant metastasis
* Life expectancy < 1 year
* Pregnancy
* Major medical illness that would preclude study treatment
* History of major wound complication or recurrent skin infection
* Known HIV positivity
* < 2 weeks elapsed from prior surgery or cytotoxic chemotherapy
* persisting acute toxicities > grade 1 in tumor-bearing limb resulting from prior treatment with anti-cancer modalities
* Cytotoxic chemotherapy, targeted therapy or investigational agents concurrent to study treatment
* Prior radiotherapy to the site of present STS.
* Chronic requirement for treatment with immuno¬suppressive agents or steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-08; Primary Completion 2019-06 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Wound Complication Rate | 3 months
  Wound Complication Rate up to 3 months after tumor resection

SECONDARY OUTCOMES:
Efficacy | 2 years
  Efficacy:
  Rate of margin-free resection Local control rate (LC) Metastasis-Free Survival (MFS) Disease-Free Survival (DFS) Disease-Specific Survival, Overall Survival (OS) Limb Preservation Rate (LP)
Safety | 2 years
  Acute toxicity as measured by CTCAE v. 4.03 Late toxicity (skin, soft tissue, joint, bone, neural toxicity) as measured by CTCAE v. 4.03
Limb Functionality | 2 years
  as measured by the Musculoskeletal Tumor Society (MSTS) rating scale and the Toronto Extremity Salvage Score (TESS)
Quality of Life | 2 years
  as measured by QLQ C30
Translational | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Röper, MD, Principal Investigator — Klinik für Strahlentherapie und Radiologische Onkologie
Locations (1):
- Klinikum rechts der Isar, Munich, Germany

REFERENCES:
- [Derived] Roper B, Heinrich C, Kehl V, Rechl H, Specht K, Wortler K, Topfer A, Molls M, Kampfer S, von Eisenharth-Rothe R, Combs SE. Study of Preoperative Radiotherapy for Sarcomas of the Extremities with Intensity-Modulation, Image-Guidance and Small Safety-margins (PREMISS). BMC Cancer. 2015 Nov 16;15:904. doi: 10.1186/s12885-015-1633-y. PMID 26573139